CLINICAL TRIAL: NCT02967263
Title: The Study of Etiology, Epidemiology and Prognostic Factors of Acute Kidney Injury
Brief Title: Etiology, Epidemiology and Prognostics of AKI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Ding Feng, professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: AKI-2016-01
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Proteinosis; Epidemiology; Risk factors
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood or urine samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hospital-acquired AKI: Adult patients with Hospital-acquired AKI

SUMMARY:
* To investigate the etiology and epidemiology of acute kidney injury (AKI).
* To find out risk factors associated with the occurence of AKI.
* To find out risk factors related to the prognosis of AKI,focusing on uremic toxins, inflammation, oxidative stress and nutritional status.
* To study on the relationship between gene polymorphism and prognosis of acute kidney injury.

DETAILED DESCRIPTION:
1. To investigate the relationship between preexisting protein-energy wasting (PEW) and adverse outcomes in patients with AKI.
2. To evaluate the association of serum nutritional variables and prognosis of AKI.
3. Given the different half-lives of serum nutritional markers, we hypothesized that the utility of serum nutritional variables as prognostic predictors may differ in early death (<7 days) and late death (>7 days, <28 days) patients.
4. To investigate the various kinds of uremic toxins in AKI, furthermore, to evaluate the relationship between uremic toxins, especially protein bound toxins, and short- or long-term mortality in AKI patients.
5. To investigate the mineral bone disorders in AKI,and to evaluate whether these markers would role as prognostic predictors of AKI.
6. Several risk factors of mortality in AKI,such as markers of PEW, inflammation and serum creatinine,have been used; however, no single indicator is considered to be a "gold standard."

ELIGIBILITY:
Inclusion Criteria:

* age >=18 years and <= 88 years
* clinically diagnosed with acute kidney injury, according KDIGO criteria.

Exclusion Criteria:

* preexisting chronic kidney failure (defined as an eGFR <60 ml/min per 1.73 m2)
* post-renal obstruction or rapid progressive glomerulonephritis as the main cause of AKI
* known acute renal dysfunction
* hospital stays <24 hours
* malignancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patients aged >18 years, with hospital-acquired acute kidney injury, from a university-affiliated hospital in Shanghai, China.
Sampling Method: Probability Sample
Enrollment: 713 (Estimated)
Dates: Start 2015-01; Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 90 days

SECONDARY OUTCOMES:
renal function survival rate | 90 days
days in hospital | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ding, PhD, Study Director — Division of Nephrology, Shanghai Ninth People's Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China